CLINICAL TRIAL: NCT06518525
Title: The Effects Of Pilates-Based Tele-Exercise On Physical And Mental Health In Primary Dysmenorrhea
Brief Title: The Effects Of Pilates-Based Tele-Exercise In Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derya Azim (Other)
Collaborators: Okan University (Other)
Responsible Party: Sponsor-Investigator, Derya Azim, Assistant Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.AYD.0.00.00
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Menstruation; Pain; Tele-Exercise; pilates
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates-based tele-exercises (Experimental): Participants in the primary dysmenorrhea study group will be given a general introduction to Pilates-based tele-exercises, and they will be taught five essential elements that they should continuously practice during the exercise process. These elements will be control, breathing, fluidity, precision, and centering. They will be instructed on how to activate the core muscles, including the transverse abdominis, pelvic floor, and multifidus muscles, through isometric contractions while exhaling (centering). The exercises will be conducted over 6 weeks, twice a week, with each session lasting 50 minutes. The exercises, predetermined by the researcher, will be performed under the supervision of a physiotherapist. Each session will be structured into warm-up exercises, main exercises, and cool-down exercises. .
  Interventions: Other: pilates-based tele-exercises
- control group (No Intervention): control group

INTERVENTIONS:
Other: pilates-based tele-exercises — pilates-based tele-exercises
  Arms: pilates-based tele-exercises

SUMMARY:
In this study, the investigators will aim to investigate the effects of Pilates-based tele-exercise on the physical and mental health of women with primary dysmenorrhea. The study will include 22 volunteers diagnosed with primary dysmenorrhea. Participants will be randomly divided into two groups. The first group will undergo Pilates-based tele-exercises (6 weeks/2 days/50 minutes) (PTTE, n=11). The second group will be a non-intervention control group (CG, n=11). Pain severity will be assessed using the Visual Analog Scale (VAS), and menstrual information will be evaluated using the Menstrual Symptom Questionnaire (MSQ), Menstrual Attitude Questionnaire (MAQ), and Functional and Emotional Dysmenorrhea Scale (FEDS). Quality of life will be assessed using the Nottingham Health Profile (NHP).

DETAILED DESCRIPTION:
In this study, the investigators will aim to investigate the effects of Pilates-based tele-exercise on the physical and mental health of women with primary dysmenorrhea. The study will include 22 volunteers diagnosed with primary dysmenorrhea. Participants will be randomly divided into two groups. The first group will undergo Pilates-based tele-exercises (6 weeks/2 days/50 minutes) (PTTE, n=11). The second group will be a non-intervention control group (CG, n=11). Pain severity will be assessed using the Visual Analog Scale (VAS), and menstrual information will be evaluated using the Menstrual Symptom Questionnaire (MSQ), Menstrual Attitude Questionnaire (MAQ), and Functional and Emotional Dysmenorrhea Scale (FEDS). Quality of life will be assessed using the Nottingham Health Profile (NHP).Inclusion criteria were determined as follows: being between 18-30 years old, diagnosed with primary dysmenorrhea during an ultrasound examination, having a PD pain score of 4-7 cm on the Visual Analog Scale (VAS), being able to attend Pilates sessions twice a week, not engaging in regular exercise, and having a regular menstrual cycle (30-35 days) and bleeding duration (3-10 days). Exclusion criteria included being pregnant, having serious comorbidities (neurological, cardiovascular, and musculoskeletal disorders), and not willing to participate in the study. Volunteers who agree to participate in the study will sign an informed consent form, after which they will be given the necessary information about the scales used in the assessment. The scales will be filled out by the participants based on their previous menstrual experiences. After the assessment, Pilates-based tele-rehabilitation exercises will be applied for 6 weeks. At the end of the 6 weeks, assessments will be repeated in both groups. The scales applied to both groups before and after the study will be uploaded to the Google Forms database and sent to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years old,
* Diagnosed with primary dysmenorrhea during an ultrasound examination,
* Having a PD pain score of 4-7 cm on the Visual Analog Scale (VAS),
* Being able to attend Pilates sessions twice a week,
* Not engaging in regular exercise,
* Having a regular menstrual cycle (30-35 days) and a bleeding duration of 3-10 days,

Exclusion Criteria:

* Being pregnant,
* Having serious comorbidities (neurological, cardiovascular, and musculoskeletal disorders),
* Not willing to participate in the study,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Sure, here is the English translation: Visual Analog Scale | Baseline and 6 weeks later
  The Visual Analog Scale (VAS) was used to assess pain in the study. The VAS is a horizontal or vertical line that is 10 cm in length. At the beginning of the line, the phrase "no pain" is placed, and at the end, "unbearable pain" is written. Participants are asked to mark the point on the line that corresponds to the severity of the pain they experience. The distance between the point where the VAS value is the lowest and the point where the patient marked is measured, and the numerical value corresponding to the pain severity is recorded
Nottingham Health Profile | Baseline and 6 weeks later
  The Nottingham Health Profile (NHP) is a quality of life assessment questionnaire developed in 1987 to determine the degree to which individuals' perceived health problems affect their daily activities. The Turkish version of the scale was developed and psychometrically evaluated by Küçükdeveci et al. The NHP consists of six sub-dimensions: pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), physical activity (8 items), and energy (3 items). The questionnaire is answered with 'yes' or 'no'. Each section of the questionnaire is calculated separately; the sub-dimension score is obtained by summing the 'yes' responses to the items in each sub-dimension and dividing by the number of items in that sub-dimension, then multiplying by 100. Each sub-dimension scores between 0 and 100, with higher scores indicating lower quality of life
Menstrual Symptom Questionnaire | Baseline and 6 weeks later
  he Menstrual Symptom Questionnaire (MSQ) was developed in English by Chesney and Tasto in 1975 to assess pain and other symptoms associated with menstruation. The Turkish validity and reliability were completed by Güvenç et al. in 2014. The scale consists of 24 items in total, in a 5-point Likert-type format. It includes three sub-dimensions: 'Negative Effects/Somatic Complaints' (13 items), 'Pain Symptoms' (6 items), and 'Coping Methods' (3 items). Participants are asked to rate the symptoms they experience during menstruation as 1 (never), 2 (rarely), 3 (sometimes), 4 (often), and 5 (always). The score for each sub-dimension is calculated as the average of the total points of the items in that sub-dimension. The total score of the MSQ is calculated by averaging the total points of all scale items; higher scores indicate greater severity of menstrual symptoms.
Menstrual Attitude Questionnaire | Baseline and 6 weeks later
  The Menstrual Attitude Questionnaire (MAQ) was developed by Brooks-Gunn and Ruble in 1980, and its validity and reliability in Turkey were established by Kulakaç et al. in 2008. The Turkish version of the MAQ consists of 33 items and five sub-scales in a Likert-type format. These sub-scales are 'Menstruation as a debilitating event' (12 items), 'Menstruation as a bothersome event' (6 items), 'Menstruation as a natural event' (5 items), 'Anticipation and prediction of menstruation' (5 items), and 'Denial of menstruation effects' (7 items). Participants are asked to select one of the following options for each question: 1. Strongly disagree, 2. Disagree, 3. Neutral, 4. Agree, and 5. Strongly agree. Higher average scores from the items, sub-dimensions, or the entire scale indicate a more positive attitude towards menstruation.
Functional and Emotional Dysmenorrhea Scale | Baseline and 6 weeks later
  The Functional and Emotional Dysmenorrhea Scale (FEDS) is used to measure functional and emotional health in dysmenorrhea. It was developed by Li et al. in 2012, and its Turkish validity and reliability were established by Gün in 2014. The FEDS consists of 14 items in total, with two sub-dimensions: functional dysmenorrhea and emotional dysmenorrhea. Participants are asked to choose the option that best describes their condition for each item: 1. Does not resemble my condition at all, 2. Does not quite resemble my condition, 3. Both resembles and does not resemble my condition, 4. Somewhat resembles my condition, 5. Very much resembles my condition. Higher scores indicate greater functional and emotional impact from dysmenorrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Atıcı, Principal Investigator — Okan University
Locations (1):
- Bandırma Onyedi Eylul University, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available for use by other researchers.